CLINICAL TRIAL: NCT06916806
Title: An Open-label, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD5492 Following Single-ascending Dose and Step-up Dose Administration to Adult Participants With Systemic Lupus Erythematosus or Idiopathic Inflammatory Myopathies or Rheumatoid Arthritis
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD5492 in Adult Participants With Systemic Lupus Erythematosus or Idiopathic Inflammatory Myopathies or Rheumatoid Arthritis.
Acronym: TITAN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9961C00001; 2024-519015-34-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-03-13; First posted 2025-04-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus; Idiopathic Inflammatory Myopathies; Rheumatoid Arthritis
Keywords: Lupus; Inflammatory Myopathy; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Muscular Diseases; Myositis; Dermatomyositis; Polymyositis; Arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis; Arthritis, Rheumatoid; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Muscular Diseases; Dermatomyositis; Polymyositis; Arthritis

STUDY DESIGN:
Intervention Model Description: Open-Label, single-arm treatment study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Single Ascending Dose with AZD5492 (Experimental): Participants will receive AZD5492 at an assigned dose as subcutaneous (SC) injection on Day 1.
  Interventions: Drug: AZD5492
- Part 2: Step-Up Dosing with AZD5492 (Experimental): Participants will receive AZD5492 as SC injection at the priming dose determined in Part 1, on Day 1, and at a target dose, based on the emergent safety data, on Day 8.
  Interventions: Drug: AZD5492

INTERVENTIONS:
Drug: AZD5492 — IMP: subcutaneous.

SUMMARY:
The purpose of this study is to measure the safety, tolerability, PK, and PD of AZD5492 administered subcutaneously in adult participants with SLE or IIM or RA

Study details include:

• The study duration will be a minimum of 180 days in addition to the screening period.

Additional follow-up visits may be required up to 12 months from study start.

* Depending on the study part they are assigned to, participants will be administered AZD5492 once (Part 1) or twice (Part 2).
* Study visits will occur at:

Screening, Days 1-4, 8, 15, 22, 30, 60, 90, 120, 150, and 180 in Part 1, Screening, Days 1-4, 8-11, 15, 22, 29, 43, 60, 90, 120, 150, and 180 in Part 2.

DETAILED DESCRIPTION:
This is an open-label, multi-centre Phase I study to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of AZD5492 in adult participants with either SLE or IIM or RA.

The study consists of 2 parts:

Part 1 - Single ascending dose (SAD) Part 1 will be a sequential SAD design in adult participants with SLE. Up to 5 dose levels of AZD5492 are planned to be investigated. Depending on emerging data, up to 4 additional dose levels may be added at the discretion of the Sponsor.

The decision to open Part 2 will be made by the Safety Review Committee (SRC) based on the evaluation of all available data including safety, tolerability, PK, and PD from Part 1 and pertinent data arising from other ongoing studies with AZD5492 will also be considered, and the dose levels and dosing strategy for Part 2 will be confirmed.

After a screening period of up to 42 days, participants will receive 1 dose of AZD5492 and be followed up for at least 179 days post-dose.

Part 2 - Step-up dosing (SUD) Part 2 will be a SUD design in adult participants who have SLE (and did not participate in Part 1), as well as adult participants with IIM or RA. In Part 2, participants will receive 2 dose administrations, 7 days apart. The first (priming) dose of the step-up regimen will be agreed by the SRC. The second (target) dose will be escalated, and a minimum of 3 target dose levels are planned to be investigated in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 70 years of age inclusive, at the time of signing the informed consent.
2. Diagnosis of SLE:

   1. Diagnosis of SLE according to the 2019 EULAR/ACR classification criteria for SLE
   2. Positive for one or more of: anti-nuclear antibodies (titre ≥ 1:80), anti-dsDNA or anti-Sm at screening.
   3. Active, moderate-severe disease at screening, defined as clinical SLEDAI-2K ≥ 4.
   4. Intolerance to, or inadequate response following at least 3 months of use to, ≥ 3 available treatments, such as the following: corticosteroids, anti-malarial drugs, calcineurin inhibitor, methotrexate, azathioprine, leflunomide, mycophenolic acid or its derivatives, cyclophosphamide, belimumab, anifrolumab, telitacicept, or B-cell depleting monoclonal antibodies.
3. Diagnosis of IIM:

   1. Must have "probable" or "definite" diagnosis of PM or DM (excluding IBM and cancer associated myositis) according to the 2017 EULAR/ACR classification criteria for adult myositis.
   2. Positive for ≥ 1 disease-specific autoantibody at screening.
   3. MMT-8 score of ≤ 142/150 and/or CDASI-A ≥ 6
   4. Fulfill at least one of the following criteria of active disease at screening:

   (i) One or more muscle enzyme elevation (CK, AST, ALT, aldolase, LDH) ≥ 1.3 × ULN (ii) If criterion 3(d)(i) is not met, then at least one of the following criteria must be met: a. Report from MRI performed within 3 months prior to screening with evidence of muscle inflammation b. Report from muscle biopsy performed within 3 months prior to screening that demonstrates active inflammation c. Report from electromyography performed within 3 months prior to screening that exhibits irritable myopathic pattern.

   (e) Intolerance or inadequate response to corticosteroids and ≥2 other SoC treatments, used for at least 3 months each, for which at least one must be a biologic SoC, immunoglobulin or cyclophosphamide.
4. Diagnosis of RA:

   (a) Diagnosis of RA as defined by the 2010 EULAR/ACR classification criteria (b) Positive for ≥ 1 disease-specific autoantibody performed by the central laboratory at screening: RF or ACPA (c) Moderate or severe disease activity defined as: (i) ≥6 tender joints and ≥6 swollen joints AND (ii) DAS28-CRP >3.2. (d) Intolerance to or inadequate response following approximately 3 month's treatment or longer to ≥2 b/tsDMARDs (with different mechanisms of action) after failing csDMARD therapy (unless csDMARD therapy is contraindicated). There is no minimum duration for taking a treatment in cases of intolerance.

Exclusion Criteria:

1. Any complications of the disease under study which are judged by the investigator to be life or organ threatening or to require treatments which are not permitted in the protocol, including but not limited to:

   1. Active severe SLE-driven renal disease.
   2. History of, or current diagnosis of, catastrophic or severe APS (for example diagnosis of an arterial or central/pulmonary venous clot) within 1 year prior to signing the ICF.
   3. Rapidly progressive and/or severe ILD or ILD that requires oxygen supplementation/therapy (of any type).
   4. Inclusion Body Myositis or cancer associated myositis.
2. Active severe, unstable or history of neuropsychiatric SLE.
3. IIM: Pulmonary function tests at screening (or within one month of screening, provided participant confirms no change in respiratory symptoms in the interim) which meet any of the following criteria:

   1. FVC ≤60% of predicted
   2. DLCO ≤70% of predicted
   3. Deterioration in either FVC or DLCO at screening compared to pulmonary function tests performed ≥3 months previously.
4. Significant history of or at risk of severe infections.
5. Participants with HIV infection.
6. Participants with evidence of chronic or active hepatitis B defined as HBsAg positive or HBcAB positive
7. Participants with evidence of chronic or active hepatitis C
8. Participants with positive COVID-19 PCR.
9. Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection.
10. Significant CNS pathology.
11. Receipt of B-cell-depleting therapy including CD19 or CD20 directed monoclonal antibodies (including but not limited to, ocrelizumab, ofatumumab, obinutuzumab, or rituximab) <3 months prior to Day 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-06-22 (Estimated); Study Completion 2027-06-22 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of AZD5492: Number of participants with treatment-emergent adverse events. | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with AEs, AESIs, and SAEs
Safety evaluation of AZD5492: Number of participants with related treatment-emergent adverse events. | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with AEs related to IMP as assessed by the investigator
Safety evaluation of AZD5492: Frequency of dose limiting toxicities (DLTs). | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with DLTs (dose-limiting toxicities) as defined in the study protocol.
Safety evaluation of AZD5492: Number of SAEs leading to death | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with SAEs leading to death.
Safety evaluation of AZD5492: Number of participants with treatment-emergent adverse events by grade. | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with AEs according ASTCT, IEC-HS, and CTCAE grades.
Tolerability evaluation of AZD5492: Number of participants with treatment-emergent vital signs abnormalities. | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with treatment-related vital signs abnormalities.
Tolerability evaluation of AZD5492: Number of participants with treatment-emergent clinical laboratory abnormalities. | Day 1 to end of the study (up to 52 weeks)
  Number and percentage of participants with treatment-related clinical laboratory abnormalities.
Tolerability evaluation of AZD5492: Number of participants with abnormal ECG. | From Day 1 up to Day 180
  Number and percentage of participants with abnormal ECG.

SECONDARY OUTCOMES:
Serum Pharmacokinetics (PK) parameters of AZD5492 (Cmax) | From Day 1 through Day 60
  Maximum observed serum drug concentration (Cmax) (μg/mL)
Serum Pharmacokinetics (PK) parameters of AZD5492 (AUC) | From Day 1 through Day 60
  Area under the serum concentration-time curve (AUC) (μg/mL*h)
Serum Pharmacokinetics (PK) parameters of AZD5492 (t1/2λz) | From Day 1 through Day 60
  Terminal elimination half-life (t1/2λz) (In hours)
Serum Pharmacokinetics (PK) parameters of AZD5492 (AUClast) | From Day 1 through Day 60
  Area under the serum concentration time curve from time zero to the time of last quantifiable analyte concentration (AUClast) (nmol*h/L)
Incidence of ADAs to AZD5492 measured in serum. | From Day 1 through Day 180
  Incidence of ADAs to AZD5492 measured in serum.
Absolute counts at Day 180 in blood CD19+ B-cells. | Day 180
  Absolute counts at Day 180 in blood CD19+ B-cells.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (3):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Iowa City, Iowa
- Canada (2):
  - Research Site, Hamilton, Ontario
  - Research Site, Sherbrooke, Quebec
- China (3):
  - Research Site, Beijing
  - Research Site, Shanghai
  - Research Site, Wuhan
- France (6):
  - Research Site, Bordeaux
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (3):
  - Research Site, Cologne
  - Research Site, Erlangen
  - Research Site, Magdeburg
- Japan (5):
  - Research Site, Bunkyō City
  - Research Site, Kita-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Kyoto
  - Research Site, Nagasaki
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Leiden
- Spain (3):
  - Research Site, Mérida
  - Research Site, Seville
  - Research Site, Valladolid
- United Kingdom (3):
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/